CLINICAL TRIAL: NCT06700954
Title: Effects of a Legume-rich Diet in the Context of the Planetary Health Diet Compared to a Western-oriented Dietary Pattern in Women and Men At Increased Risk of Cardiovascular and Neurodegenerative Diseases
Brief Title: Effects of a Legume-rich Diet in the Context of the Planetary Health Diet Compared to a Western-oriented Dietary Pattern in Participants with Increased Cardiometabolic Risk
Acronym: LeguPlan_2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: Federal Ministry of Food and Agriculture (BMEL) (Unknown); Federal Office of Agriculture and Food (BLE) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Prof. Dr. Sarah Egert, University of Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BMEL: 2822EPS008 2
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- legume-rich Planetary Health Diet (Experimental): legume-rich diet based on the Planetary Health Diet, with a focus on vegetable protein
  Interventions: Other: legume-rich Planetary Health Diet
- control diet based on Western Diet low in legumes (Experimental): diet based on the Western dietary pattern including animal protein sources (= control diet)
  Interventions: Other: control diet based on Western Diet low in legumes

INTERVENTIONS:
Other: legume-rich Planetary Health Diet — legume-rich diet based on the Planetary Health Diet, with a focus on vegetable protein
  Arms: legume-rich Planetary Health Diet
Other: control diet based on Western Diet low in legumes — diet based on the Western dietary pattern including animal protein sources (= control diet)
  Arms: control diet based on Western Diet low in legumes

SUMMARY:
The aim of the study is to systematically investigate the effects of a diet enriched with legumes in a dietary pattern approach (Planetary Health Diet) compared to a control diet low in legumes in older people with a risk phenotype for cardiovascular and neurodegenerative diseases. For this purpose, a controlled, six-week nutritional intervention study will be carried out in a parallel design. A total of 100 subjects (aged 50 - 75 years) will be randomly assigned to one of two intervention groups: i) a legume-rich diet based on the Planetary Health Diet, with a focus on plant protein, ii) a diet based on the Western dietary pattern including animal protein sources (= control diet). The target variables include parameters of lipid, glucose and insulin metabolism as well as biomarkers of inflammation and endothelial activation, proteomics and neurodegeneration markers. Furthermore, pulse wave velocity is measured to assess vascular function and neuropsychological target variables (e.g. hunger, satiety) are recorded using questionnaires.

DETAILED DESCRIPTION:
The aim of the study is to systematically investigate the effects of a diet enriched with legumes in the dietary pattern approach (Planetary Health Diet) compared to a control diet low in legumes in older people with a risk phenotype for cardiovascular and neurodegenerative diseases. For this purpose, a controlled, six-week nutritional intervention study will be carried out in a parallel design. A total of 100 subjects (aged 50 - 75 years) will be randomly assigned to one of two intervention groups: i) a legume-rich diet based on the Planetary Health Diet, with a focus on plant protein, ii) a diet based on the Western dietary pattern including animal protein sources (= control diet). The target variables include parameters of lipid, glucose and insulin metabolism as well as biomarkers of inflammation and endothelial activation, proteomics and neurodegeneration markers. Furthermore, pulse wave velocity is measured to assess vascular function and neuropsychological target variables (e.g. hunger, satiety) are recorded using questionnaires. The subjects come to the study center for examination before the start of the intervention (visit 1), after three weeks (mid-intervention, visit 2) and after six weeks (end of intervention, visit 3).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Non-smoking
* BMI: 27 - 34,9 kg/m2
* Waist circumference (women ≥ 80 cm, men ≥ 94 cm)
* Systolic blood pressure: ≥ 120 mmHg, diastolic blood pressure: ≥ 80 mmHg
* At least one of the following criteria:
* Fasting triglycerides in serum: ≥ 150 mg/dL
* Fasting LDL cholesterol in serum ≥160 mg/dL
* Fasting HDL-Cholesterol in serum: women < 50 mg/dl, men < 40 mg/dL
* Fasting glucose in plasma: ≥ 100 mg/dL
* CRP in serum 0,2-3 mg/dL

Exclusion Criteria:

* food intolerances and allergies (especially legumes)
* Smoking
* malabsorption syndromes
* thyroid diseases
* impaired renal function
* chronic liver disease
* heart failure
* myocardial infarction
* insulin-dependent diabetes mellitus
* chronic inflammatory diseases
* tumors
* anemia
* immunosuppression
* intake of supplements (e.g., fish oil)
* Participation in another study
* other exclusion criteria at the discretion of the physician/ investigator

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pameters of glucose metabolism in blood | postprandial period of 2 hours (t = 0,2) in week 1 and week 6 of intervention
  Glucose (mg/dL)

SECONDARY OUTCOMES:
Parameters of glucose metabolism in blood | postprandial period of 2 hours (t = 0,2) in week 1 and week 6 of intervention
  Insulin (nmol/L)
Parameters of glucose metabolism in blood | postprandial period of 2 hours (t = 0,2) in week 1 and week 6 of intervention
  GLP-1 (pg/mL)
Parameters of glucose metabolism in blood | postprandial period of 2 hours (t = 0,2) in week 1 and week 6 of intervention
  Glucagon (pg/mL)
Parameters of glucose metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  HbA1c (%)
Parameters of glucose metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Fructosamine (µmol/l)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Triglycerides (mg/dL)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Total cholesterol (mg/dL)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  LDL cholesterol (mg/dL)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  HDL cholesterol (mg/dL)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Free fatty acids (mmol/L)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Lipoprotein(a) (mg/dL/nmol/L)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Apo A1 (g/L)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Apo B (g/L)
Parameters of lipid metabolism in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Fatty acid composition of serum phospholipids
Blood urea | Fasting (t=0) in week 1 and week 6 of intervention
  Urea in blood (mg/dL)
Uric acid in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Uric acid in blood (mg/dL)
Parameters of endothelial function in blood | Fasting (t=0) in week 1 and week 6 of intervention
  ADMA (µmo/L)
Parameters of inflammation in blood | Fasting (t=0) in week 1 and week 6 of intervention
  IL-6 (pg/mL)
Parameters of Hunger and Satiety in blood | Fasting (t=0) in week 1 and week 6 of intervention
  Ghrelin (pg/mL)
Endothelial function | Fasting (t=0) in week 1 and week 6 of intervention
  pulse wave velocity (m/s) with the vicorder device
Liver enzymes | Fasting (t=0) in week 1 and week 6 of intervention
  GGT (U/L)
Liver enzymes | Fasting (t=0) in week 1 and week 6 of intervention
  ALT (U/L)
Liver enzymes | Fasting (t=0) in week 1 and week 6 of intervention
  AST (U/L)
Small blood count | Fasting (t=0) in week 1 and week 6 of intervention
Ferritin | Fasting (t=0) in week 1 and week 6 of intervention
  Ferritin (µg/L)
Adiponectin | Fasting (t=0) in week 1 and week 6 of intervention
  Adiponectin (µg/ml)
Parameters oft the antioxidant system | Fasting (t=0) in week 1 and week 6 of intervention
  vitamin C
Parameters oft the antioxidant system | Fasting (t=0) in week 1 and week 6 of intervention
  vitamin E
Parameters oft the antioxidant system | Fasting (t=0) in week 1 and week 6 of intervention
  ß-carotine
Parameters oft the antioxidant system | Fasting (t=0) in week 1 and week 6 of intervention
  B vitamins
trace elements | Fasting (t=0) in week 1 and week 6 of intervention
  iron
trace elements | Fasting (t=0) in week 1 and week 6 of intervention
  cupper
trace elements | Fasting (t=0) in week 1 and week 6 of intervention
  zinc
trace elements | Fasting (t=0) in week 1 and week 6 of intervention
  selen
Proteomics | Fasting (t=0) in week 1 and week 6 of intervention
Neurodegenerative markers | Fasting (t=0) in week 1 and week 6 of intervention
  GFAP
Neurodegenerative markers | Fasting (t=0) in week 1 and week 6 of intervention
  Aβ42
Neurodegenerative markers | Fasting (t=0) in week 1 and week 6 of intervention
  Aβ40
Neurodegenerative markers | Fasting (t=0) in week 1 and week 6 of intervention
  NF-L
Blood pressure | Fasting (t=0) in week 1 and week 6 of intervention
  Blood pressure (mmHg)
REE | Fasting (t=0) in week 1 and week 6 of intervention
  REE (kcal/24h)
Anthropometic measurements | Fasting (t=0) in week 1 and week 6 of intervention
  weight (kg)
Anthropometic measurements | Fasting (t=0) in week 1 and week 6 of intervention
  fat mass (%)
Anthropometic measurements | Fasting (t=0) in week 1 and week 6 of intervention
  waist circumference (cm)
Neuropsychological parameters | Fasting (t=0) in week 1 and week 6 of intervention
  Assessment of memory via a validated neuropsychological questionaire (paper pencil, e.g. higher reproduction of memorised visual and verbal information = better memory; visual part: maximum points: 31 = all visual information memorised, minimum points: 0 = no visual information memorised; verbal part: maximum points: 24 = all verbal information memorised, minimum points: 0 = no verbal information memorised)
Fecal fatty acid profile | Fasting (t=0) in week 1 and week 6 of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutritional and Food Sciences, Nutrition Physiology, Bonn, North Rhine-Westphalia, Germany